CLINICAL TRIAL: NCT05784051
Title: Prophylactic Frequent Premature Ventricular complexeS sUPPression on Left ventriculaR Function impairmEnt in aSymptomatic patientS
Acronym: SUPPRESS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP180618
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Premature Ventricular Contractions; Ventricular Dysfunction, Left
MeSH Terms: conditions — Ventricular Premature Complexes; Ventricular Dysfunction, Left | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The SUPPRESS study will be a national multicenter randomized open label trial using the PROBE study design (Prospective Randomized Open Blinded End-point).
  Patients fulfilling the inclusion criteria (asymptomatic patients with frequent (> 10%/day) PVCs and normal LVEF) and without any exclusion criteria that agree to enter the protocol will be randomized to:
  1. Experimental group: 149 patients treated for PVCs with drug therapy and/or catheter ablation/ medical treatment including drug administration ± catheter ablation (Ablation can be performed if the PVC burden remain >10% after 2 lines of AAD treatment).
  2. Control group: 149 patients with therapeutic abstention or no treatment modification such as drug therapy/ Therapeutic abstention or no modification of therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients treated for PVCs with drug therapy and/or catheter ablation/ medical treatment including drug administration ± catheter ablation (Ablation can be performed if the PVC burden remain >10% after 2 lines of AAD treatment).
  Interventions: Drug: Experimental group
- Control group (Active Comparator): Patients with therapeutic abstention or no treatment modification such as drug therapy/ Therapeutic abstention or no modification of therapy
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: Experimental group — medical treatment including drug administration ± catheter ablation (Ablation can be performed if the PVC burden remain >10% after 2 lines of AAD treatment).
  Other Names: medical treatment
  Arms: Experimental group
Drug: Control group — patients of this group have no therapeutic or no treatment modification such as drug therapy
  Other Names: Therapeutic abstention or no modification of therapy
  Arms: Control group

SUMMARY:
The main objective of the study is to demonstrate that prophylactic treatment of patients with asymptomatic frequent (>10%) PVCs is superior to simple follow-up strategy with no therapy to prevent subsequent LV dysfunction at 24 months. The prophylactic treatment is based on drugs ± ablation (ablation can be performed if the PVC burden remain >10% after 2 lines of AAD treatment since the initiation of the study).

The primary endpoint will be the development of LV dysfunction (PVC-iCMP) defined as a 15% relative LVEF decrease (and/or a LVEF <50%) within 2 years following randomization, on cardiac magnetic resonance imaging (cMRI) (or transthoracic echocardiography (TTE) when not possible).

DETAILED DESCRIPTION:
Premature ventricular contractions (PVCs) are frequently encountered in clinical practice, in the setting of underlying heart disease as well as in "normal" hearts. Frequent PVCs have been shown to impact long term prognosis in patients with structurally normal hearts,[1] as well as in documented cardiomyopathy. In both settings, PVCs may cause symptoms and, in rare cases, sudden cardiac death. For about two decades, it has been accepted that frequent PVCs may also induce left ventricular (LV) dysfunction called PVC-induced cardiomyopathy (PVC-iCMP). Indeed, PVC suppression by using drugs or catheter ablation has been associated with full recovery of left ventricular dysfunction.[2-4] De facto, PVC-iCMP diagnosis as well as identification of predictors has always been established retrospectively. Therefore, risk stratification or simply knowing the exact incidence of the disease in exposed patients remain difficult.

European and US guidelines recommend to treat symptomatic PVC patients regardless of the burden or their risk profile, as well as "frequent PVCs" associated with LV dysfunction (Experts tend to consider worthwhile treating for burden >10%, which was the lowest burden associated with PVC-iCMP).

However, there is no clear recommendation for asymptomatic patients exposed to very frequent PVCs, at risk of developing cardiomyopathy. As no previous studies included such population, expert suggested that these patients should be at least closely followed. Consequently, management of such patients is widely heterogeneous.

The hypothesis of this study is that prophylactic suppression of very frequent PVCs (>10%) will prevent or significantly reduce the incidence of PVC-iCMP.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria (all must be present):

1. 18 ≤ Age ≤ 85
2. PVC burden ≥ to 10% regardless of current or preexisting antiarrhythmic drug intake (for instance, a patient under betablocker therapy because of his PVCs or hypertension can be included)
3. Asymptomatic status
4. Normal (>or= 55%) LVEF. Patients with underlying cardiomyopathy can be included as long as LV function remains preserved.
5. Signed informed consent

Exclusion criteria (any of them):

1. Pregnant woman or Female of childbearing potential without effective method of birth control or nursing woman.
2. Patients that can't undergo MRI study
3. De novo requirement for antiarrhythmic drug prescription for another indication (e.g. atrial fibrillation…)
4. The physician already decided that the patient requires drug initiation or escalation;
5. Ischemic cardiomyopathy requiring revascularization (PCI or surgery)
6. History of LV dysfunction
7. Participation in another research involving the human person
8. Patient under legal protection
9. Non affiliation to a social security scheme

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
occurence of Left ventricular dysfunction (PVC-iCMP) | 24 months
  The primary endpoint will be the development of left ventricular dysfunction (PVC-iCMP) defined as a 15% relative LVEF decrease (and/or a LVEF <50%) within 2 years following randomization, on cardiac magnetic resonance imaging (cMRI) (or transthoracic echocardiography (TTE) when not possible).

SECONDARY OUTCOMES:
Rate of Death | 24 months
  Death from any cause
Rate of Cardiovascular Death | 24 months
  measure of safety endpoint: Death cause of death
Rate of Hospitalization for an adverse event | 24 months
  occurence of adverse events (AE) and serious adverse events (SAE) within follow-up that may be linked or not to anti-arrhythmic drugs (AAD) or ablation procedure
Percentage of patients with a PVC burden <10% | during 24 months follow up
  measure of efficacy endpoints:
  PVC burden will be measured the second year following randomization
LVEF variation | 24 months
  LVEF variation(from baseline to M24)
Nt-ProBNP relative variation | 24 months
  Nt-ProBNP relative variation from baseline to M24

IPD SHARING:
Plan to Share IPD: No